CLINICAL TRIAL: NCT02908074
Title: A 6 Month, Double-blind Safety Extension Study of MBGS205
Brief Title: A 6 Month Safety Extension Study of MBGS205
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mereo BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MBGS206
Record Dates: First submitted 2016-09-12; First posted 2016-09-20 (Estimated); Results first posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-04

CONDITIONS: Hypogonadotropic Hypogonadism
Keywords: Hypogonadotropic; hypogonadism; testosterone
MeSH Terms: conditions — Hypogonadism | interventions — leflutrozole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BGS649 0.1 mg (Experimental): Drug: BGS649 Dose 1 weekly
  Interventions: Drug: BGS649
- BGS649 0.3 mg (Experimental): Drug: BGS649 Dose 2 weekly
  Interventions: Drug: BGS649
- BGS649 1.0 mg (Experimental): Drug: BGS649 Dose 3 weekly
  Interventions: Drug: BGS649

INTERVENTIONS:
Drug: BGS649 — Capsules will be taken weekly for a maximum of 24 weeks
  Other Names: Leflutrozole

SUMMARY:
Phase IIb, multicentre, double-blind, randomised, placebo-controlled parallel-group 36-week study evaluating safety and efficacy of BGS649 in male obese subjects with hypogonadotropic hypogonadism (HH)

DETAILED DESCRIPTION:
This is a 6 months, active treatment, extension study, open to subjects who have completed full 24 weeks in Study MBGS205 (A Phase IIb multicentre, double-blind, dose-ranging, randomised, placebo-controlled study evaluating safety and efficacy of BGS649 in male obese subjects with hypogonadotropic hypogonadism [HH]).The main purpose of Study MBGS206 is to evaluate long term safety and efficacy parameters in subjects after 12 months exposure with BGS649.

ELIGIBILITY:
Inclusion Criteria:

* Participating in Study MBGS205 and completion of the 24 week treatment period without meeting any discontinuation criteria of Study MBGS205
* In opinion of the investigator has been compliant with the requirements of the Study MBGS205 protocol.

Exclusion Criteria:

-Meeting any of the discontinuation criteria of initial Study MBGS205

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2018-09-08 (Actual); Study Completion 2018-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Jones, Principal Investigator — Barnsley Hospital NHS Foundation Trust
Locations (37):
- United States (37):
  - Mereo Research Site, Mobile, Alabama
  - Mereo Research Site, Chandler, Arizona
  - Mereo Research Site, Phoenix, Arizona
  - Mereo Research Site, Scottsdale, Arizona
  - Mereo Research Site, Anaheim, California
  - Mereo Research Site, Greenbrae, California
  - Mereo Research Site, Lincoln, California
  - Mereo Research Site, Los Angeles, California
  - Mereo Research Site, San Diego, California
  - Mereo Research Site, Bradenton, Florida
  - Mereo Research Site, DeLand, Florida
  - Mereo Research Site, Fort Myers, Florida
  - Mereo Research Site, Hialeah, Florida
  - Mereo Research Site, St. Petersburg, Florida
  - Mereo Research Site, Meridian, Idaho
  - Mereo Research Site, Evansville, Indiana
  - Mereo Research Site, Marrero, Louisiana
  - Mereo Research Site, Elkridge, Maryland
  - Mereo Research Site, Henderson, Nevada
  - Mereo Research Site, Las Vegas, Nevada
  - Mereo Research Site, Albany, New York
  - Mereo Research Site, Garden City, New York
  - Mereo Research Site, Great Neck, New York
  - Mereo Research Site, New York, New York
  - Mereo Research Site, Rochester, New York
  - Mereo Research Site, Charlotte, North Carolina
  - Mereo Research Site, Raleigh, North Carolina
  - Mereo Research Site, Winston-Salem, North Carolina
  - Mereo Research Site, Mt. Pleasant, South Carolina
  - Mereo Research Site, Nashville, Tennessee
  - Mereo Research Site, Dallas, Texas
  - Mereo Research Site, Fort Worth, Texas
  - Mereo Research Site, Pearland, Texas
  - Mereo Research Site, San Antonio, Texas
  - Mereo Research Site, West Jordan, Utah
  - Mereo Research Site, Norfolk, Virginia
  - Mereo Research Site, Kenosha, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants receiving active doses of BGS649 in Study MBGS205 continued with the same dose in Study MBGS206; Participants receiving placebo in Study MBGS205 were re-randomised at the Baseline visit to receive one of the 3 treatment regimens (BGS649 0.1 mg, 0.3 mg, and 1.0 mg) in a 1:1:1 ratio, and were only assessed for safety in study MBGS206.
Groups:
- Placebo to BGS649 0.1 mg: Drug: BGS649 Dose 1 weekly
  BGS649: Capsules will be taken weekly for a maximum of 24 weeks
- Placebo to BGS649 0.3 mg: Drug: BGS649 Dose 2 weekly
  BGS649: Capsules will be taken weekly for a maximum of 24 weeks
- Placebo to BGS649 1.0 mg: Drug: BGS649 Dose 3 weekly
  BGS649: Capsules will be taken weekly for a maximum of 24 weeks
Period: Overall Study
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg | Placebo to BGS649 0.1 mg | Placebo to BGS649 0.3 mg | Placebo to BGS649 1.0 mg
Started | 38 | 33 | 31 | 13 | 17 | 11
Received at Least 1 Dose of Study Drug | 38 | 33 | 30 | 13 | 17 | 10
Safety Population | 38 | 33 | 30 | 13 | 17 | 10
Intention-to-treat (ITT) Population | 38 | 33 | 30 | 0 | 0 | 0
Completed | 29 | 27 | 25 | 10 | 13 | 7
Not Completed | 9 | 6 | 6 | 3 | 4 | 4
Not completed — sponsor/ICON decision | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 5 | 2 | 0 | 0 | 1 | 0
Not completed — AESI | 1 | 0 | 1 | 0 | 1 | 0
Not completed — Discontinuation criteria per protocol | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 2 | 2 | 2 | 2 | 2
Not completed — Lost to Follow-up | 0 | 1 | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received at least 1 administration of the study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg | Placebo to BGS649 0.1 mg | Placebo to BGS649 0.3 mg | Placebo to BGS649 1.0 mg | Total
Number analyzed (Participants) | 38 | 33 | 30 | 13 | 17 | 10 | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (7.34) | 51.9 (7.76) | 50.0 (9.98) | 48.9 (11.04) | 49.8 (8.93) | 51.1 (8.32) | 51.0 (8.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 38 | 33 | 30 | 13 | 17 | 10 | 141
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 8 | 9 | 1 | 1 | 2 | 29
  White | 30 | 23 | 19 | 11 | 15 | 8 | 106
  More than one race | 0 | 2 | 0 | 1 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Bone Mineral Density Measured by DEXA (g/cm^2) From Baseline in Study MBGS205 to Week 48 in Study MBGS206
Description: Percentage change in lumbar bone mineral density measured by DEXA (g/cm^2) from Baseline in Study MBGS205 to Week 48 in Study MBGS206 by dose group in participants randomised to active treatment in MBGS205.
Time Frame: At 48 weeks compared to baseline in MBGS205
Population: The Intention-to-treat (ITT) population included all participants who: were randomised, and received at least 1 dose of study medication, and provided a Baseline lumbar spine bone mineral density (BMD) measure in MBGS205 and at least one available evaluation of lumbar spine post-Baseline in MBGS206. Here, the "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage change
Groups:
- BGS649 0.1 mg: Drug: BGS649 Dose 1 weekly
  BGS649: Capsules will be taken weekly for a maximum of 24 weeks in MBGS205 and 24 weeks in MBGS206
- BGS649 0.3 mg: Drug: BGS649 Dose 2 weekly
  BGS649: Capsules will be taken weekly for a maximum of 24 weeks in MBGS205 and 24 weeks in MBGS206
- BGS649 1.0 mg: Drug: BGS649 Dose 3 weekly
  BGS649: Capsules will be taken weekly for a maximum of 24 weeks in MBGS205 and 24 weeks in MBGS206
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg
Number analyzed (Participants) | 21 | 16 | 16
Percentage change | -2.24 (3.157) | -3.31 (5.301) | -1.68 (3.095)

2. Secondary Outcome: Percentage Change From Baseline in DEXA Scan Density (g/cm^2) by Location for Subjects Randomised to Active Treatment in Study MBGS205 (Over-read)
Description: Percentage change from baseline in hip (total and femoral neck) bone mineral density measured by DEXA (g/cm^2) from Baseline in Study MBGS205 to Week 48 in Study MBGS206
Time Frame: 48 Weeks
Population: The ITT population included all participants who: were randomised, and received at least 1 dose of study medication, and provided a Baseline lumbar spine BMD measure in MBGS205 and at least one available evaluation of lumbar spine post-Baseline in MBGS206. Here, the "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg
Number analyzed (Participants) | 24 | 17 | 17
percentage of change
  Bone Density (Hip) | 0.01 (3.407) | -1.71 (3.590) | 0.61 (4.304)
  Bone Density (Femoral Neck) | -1.09 (5.205) | -2.60 (6.899) | -0.15 (5.155)
  Bone Density (Lumbar Spine) | -1.94 (3.378) | -3.31 (5.301) | -1.99 (3.159)

3. Secondary Outcome: Descriptive Summary of Percentage Change in Bone Turnover Markers for Subjects Randomised to Active Treatment in Study MBGS205
Description: Percentage change from baseline in bone turnover markers (C-terminal telopeptide [CTx1], osteocalcin, bone alkaline phosphatase, and procollagen type 1 N-propeptide [P1NP]) from Baseline in Study MBGS205 to Week 48 in Study MBGS206
Time Frame: 48 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg
Number analyzed (Participants) | 28 | 26 | 23
ug/L
  2Type I Collagen C-Telopeptides | 83.28 (164.647) | 64.42 (64.473) | 57.91 (82.289)
  Procollagen 1 N-Terminal Propeptide | 40.40 (32.108) | 37.62 (44.742) | 34.17 (35.017)
  Osteocalcin | 13.79 (17.525) | 18.86 (28.545) | 15.28 (25.980)

4. Secondary Outcome: Percentage of Subjects With DEXA Scan T-score ≤ -2.5 at Week 48 by Location
Description: Proportion of subjects with DEXA scan T- scores ≤ -2.5 at Week 48 in MBGS206 compared to baseline in MBGS205 by body location (using overread scan images).
Time Frame: 48 Weeks
Population: The ITT population included all participants who: were randomised, and received at least 1 dose of study medication, and provided a Baseline lumbar spine BMD measure in MBGS205 and at least one available evaluation of lumbar spine post-Baseline in MBGS206. Here, the "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure and "Number analyzed" is the number of participants evaluated for each location.
Measure: Count of Participants; unit: Participants
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg | Placebo to BGS649 0.1 mg | Placebo to BGS649 0.3 mg | Placebo to BGS649 1.0 mg
Number analyzed (Participants) | 24 | 17 | 16 | 8 | 13 | 4
Participants
  T - Score (Hip) ≤ -2.5: number analyzed (Participants) | 24 | 17 | 16 | 8 | 13 | 3
  T - Score (Hip) ≤ -2.5 | 0 | 0 | 0 | 0 | 0 | 0
  T - Score (Femoral Neck) ≤ -2.5: number analyzed (Participants) | 24 | 17 | 16 | 8 | 13 | 3
  T - Score (Femoral Neck) ≤ -2.5 | 0 | 0 | 0 | 0 | 0 | 0
  T - Score (Lumbar Spine) ≤ -2.5: number analyzed (Participants) | 22 | 17 | 16 | 8 | 13 | 4
  T - Score (Lumbar Spine) ≤ -2.5 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Percentage Change From Baseline in Bone Mineral Density by Location and Vitamin D Deficiency
Description: Percentage change from baseline in bone density and bone biomarkers for vitamin D deficiency from Baseline in Study MBGS205 to Week 48 in Study MBGS206. Bone mineral density (g/cm^2) measured by DEXA over-read by a central reader.
Time Frame: 48 Weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage change from baseline in DEXA
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg | Placebo to BGS649 0.1 mg | Placebo to BGS649 0.3 mg | Placebo to BGS649 1.0 mg
Number analyzed (Participants) | 17 | 13 | 14 | 6 | 8 | 2
percentage change from baseline in DEXA
  Bone Density (Hip) (g/cm2): number analyzed (Participants) | 17 | 13 | 13 | 6 | 7 | 1
  Bone Density (Hip) (g/cm2) | -0.86 (3.129) | -1.81 (3.684) | 1.22 (4.532) | -0.78 (3.910) | 0.09 (1.497) | 4.36 (NA) — SD not calculable for single participant
  Bone Density (Femoral Neck) (g/cm2): number analyzed (Participants) | 17 | 13 | 13 | 6 | 7 | 2
  Bone Density (Femoral Neck) (g/cm2) | -1.93 (5.743) | -2.27 (6.739) | 0.19 (5.161) | -0.56 (4.485) | 0.16 (2.640) | 3.02 (NA) — SD not calculable for single participant
  Bone Density (Lumbar Spine) (g/cm2): number analyzed (Participants) | 16 | 12 | 14 | 6 | 8 | 2
  Bone Density (Lumbar Spine) (g/cm2) | -2.10 (3.623) | -3.86 (5.966) | -2.01 (3.520) | 1.54 (4.463) | -0.08 (2.017) | -3.12 (1.691)

6. Secondary Outcome: Change From Baseline of Oestradiol (Absolute) From Baseline in Study MBGS205 to Week 48
Description: Descriptive Summary of Oestradiol and Testosterone/Oestradiol Ratio for Subjects Randomised to Active Treatment in Study MBGS205
Time Frame: 48 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Oestradiol (pg/mL)
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg
Number analyzed (Participants) | 28 | 27 | 24
Oestradiol (pg/mL) | -12.750 (13.4264) | -11.852 (5.6820) | -12.917 (9.0117)

7. Secondary Outcome: Change From Baseline of Oestradiol (Percentage) From Baseline in Study MBGS205 to Week 48
Description: Descriptive Summary of Percentage Change in Oestradiol and Testosterone/Oestradiol Ratio for Subjects Randomised to Active Treatment in Study MBGS205
Time Frame: 48 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage from baseline at Week 48
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg
Number analyzed (Participants) | 28 | 27 | 24
percentage from baseline at Week 48 | -39.54 (33.295) | -47.00 (17.852) | -48.30 (19.752)

8. Secondary Outcome: Analysis of Proportion of Subjects That Overshoot Testosterone for Subjects Randomised to Active Treatment in Study MBGS205
Description: Proportion of subjects that overshoot testosterone (total testosterone above 1000 ng/dl [35 nmol/L], from first dose of study drug in Study MBGS205 until study completion)
Time Frame: 48 Weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg
Number analyzed (Participants) | 25 | 17 | 21
Participants | 0 | 0 | 2

9. Secondary Outcome: Change From Baseline in PSA From Baseline in Study MBGS205 to Week 48 in Study MBGS206
Description: Summary of Laboratory Test Results and Change from Baseline: PSA for Subjects Randomised to Active Treatment in Study MBGS205
Time Frame: 48 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Prostate Specific Antigen (ug/L)
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg
Number analyzed (Participants) | 28 | 27 | 24
Prostate Specific Antigen (ug/L) | 0.163 (0.2454) | 0.164 (0.6410) | 0.169 (0.6246)

10. Secondary Outcome: Change From Baseline in Haematocrit at Week 48
Description: Change from baseline in haematocrit from Baseline in Study MBGS205 to Week 48 in Study MBGS206
Time Frame: 48 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: RATIO (Change)
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg
Number analyzed (Participants) | 28 | 27 | 24
RATIO (Change) | 0.0128 (0.02273) | 0.0136 (0.02517) | 0.0286 (0.03410)

11. Secondary Outcome: Change From Baseline in Blood Pressure From Baseline to Week 48MBGS205
Description: Change from baseline in blood pressure (systolic and diastolic measured in mmHg) Baseline in Study MBGS205 to Week 48 in Study MBGS206.
Time Frame: 48 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Blood Pressure (mmHg) (Change)
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg
Number analyzed (Participants) | 20 | 17 | 19
Blood Pressure (mmHg) (Change)
  Systolic Blood Pressure | 2.7 (7.13) | 2.6 (12.64) | -0.7 (8.34)
  Diastolic Blood Pressure | -0.2 (8.12) | 1.1 (4.41) | 1.6 (8.30)

12. Secondary Outcome: Percentage of Subjects Achieving Normalisation of Bioavailable (Total) Testosterone at Wk 48
Description: Percentage of subjects where bioavailable testosterone was normalised at week 48 in Study MBGS206. Where normalisation was considered testosterone in the range 300-1000 mg/dL.
Time Frame: 48 Weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg | Placebo to BGS649 0.1 mg | Placebo to BGS649 0.3 mg | Placebo to BGS649 1.0 mg
Number analyzed (Participants) | 25 | 17 | 21 | 8 | 11 | 5
Participants | 25 | 17 | 19 | 6 | 11 | 5

13. Secondary Outcome: Descriptive Summary of Total Testosterone (ng/dL) for Subjects Randomised to Active Treatment in Study MBGS205
Description: Change from baseline in total, free and bioavailable testosterone from Baseline in Study MBGS205 to Week 48 in Study MBGS206
Time Frame: 48 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Total Testosterone (ng/dL) Change
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg
Number analyzed (Participants) | 20 | 16 | 17
Total Testosterone (ng/dL) Change | 241.0 (99.14) | 290.6 (109.64) | 378.9 (158.67)

14. Secondary Outcome: Change From Baseline in Free and Bioavailable Testosterone
Description: Change from baseline in free and bioavailable (total) testosterone from baseline in Study MBGS205 to Week 48 in Study MBGS206.
Time Frame: 48 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: (ng/dL) and (ng/L), respectively
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg | Placebo to BGS649 0.1 mg | Placebo to BGS649 0.3 mg | Placebo to BGS649 1.0 mg
Number analyzed (Participants) | 20 | 16 | 17 | 7 | 11 | 3
(ng/dL) and (ng/L), respectively
  Bioavailable Testosterone (ng/dL) | 162.12 (70.686) | 191.23 (76.431) | 255.57 (103.758) | 168.71 (111.634) | 240.25 (111.842) | 255.27 (111.674)
  Testosterone, Free (ng/L) | 60.28 (25.020) | 72.65 (26.674) | 94.82 (35.674) | 61.01 (40.632) | 84.62 (38.353) | 90.47 (37.064)

15. Secondary Outcome: Change From Baseline in Luteinizing Hormone From Baseline to Week 48
Description: Change from baseline of LH from Baseline in Study MBGS205 to Week 48 in Study MBGS206.
Time Frame: 48 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Luteinizing Hormone (mIU/mL)
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg | Placebo to BGS649 0.1 mg | Placebo to BGS649 0.3 mg | Placebo to BGS649 1.0 mg
Number analyzed (Participants) | 20 | 17 | 19 | 7 | 11 | 3
Luteinizing Hormone (mIU/mL) | 2.683 (1.6586) | 3.665 (2.3477) | 3.613 (2.7807) | 3.973 (4.1420) | 4.834 (3.1930) | 2.720 (0.5071)

16. Secondary Outcome: Change From Baseline in Follicle Stimulating Hormone at Week 48
Description: Change from Baseline in Study MBGS205 to Week 48 in Study MBGS206 in follicle stimulating hormone (FSH).
Time Frame: 48 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Follicle Stimulating Hormone (mIU/mL)
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg
Number analyzed (Participants) | 20 | 17 | 19
Follicle Stimulating Hormone (mIU/mL) | 5.473 (2.9494) | 7.509 (3.0235) | 6.781 (5.2389)

17. Secondary Outcome: Percentage Change in Bone Alkaline Phosphatase
Description: Percentage change in baseline in alkaline phosphatase from baseline in study MBGS205 to week 48 in MBGS206.
Time Frame: 48 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg | Placebo to BGS649 0.1 mg | Placebo to BGS649 0.3 mg | Placebo to BGS649 1.0 mg
Number analyzed (Participants) | 28 | 26 | 23 | 10 | 13 | 6
U/L | 12.67 (16.025) | 3.85 (17.856) | 15.28 (5.82) | 14.46 (22.493) | -3.40 (16.672) | 3.80 (13.025)

ADVERSE EVENTS:
Time Frame: Overall Adverse Events During the Active Treatment Period and Follow-up (48 Week Treatment Period plus 12 Weeks follow-up)
Description: The safety population included all participants who received at least 1 administration of the study medication.
Arm/Group | BGS649 0.1 mg | BGS649 0.3 mg | BGS649 1.0 mg | Placebo to BGS649 0.1 mg | Placebo to BGS649 0.3 mg | Placebo to BGS649 1.0 mg
All-Cause Mortality (participants affected / at risk) | 0/38 | 1/33 | 0/30 | 0/13 | 0/17 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/38 | 2/33 | 1/30 | 0/13 | 0/17 | 0/10
Other Adverse Events (participants affected / at risk) | 27/38 | 23/33 | 25/30 | 10/13 | 12/17 | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BGS649 0.1 mg (N=38) | BGS649 0.3 mg (N=33) | BGS649 1.0 mg (N=30) | Placebo to BGS649 0.1 mg (N=13) | Placebo to BGS649 0.3 mg (N=17) | Placebo to BGS649 1.0 mg (N=10)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BGS649 0.1 mg (N=38) | BGS649 0.3 mg (N=33) | BGS649 1.0 mg (N=30) | Placebo to BGS649 0.1 mg (N=13) | Placebo to BGS649 0.3 mg (N=17) | Placebo to BGS649 1.0 mg (N=10)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1) | 4 (5) | 2 (2) | 5 (6) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatic specific antigen increased (Investigations) | 5 (6) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Haematocrit increased (Investigations) | 3 (6) | 1 (3) | 2 (2) | 0 (0) | 1 (3) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Antinuclear antibody positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Red blood cells urine positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast enlargement (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testicular hypertrophy (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Penis disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spontaneous penile erection (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (7) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thoracic outlet syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fascial rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Libido decreased (Psychiatric disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Apathy (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polycythaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperadrenalism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-03-28): https://cdn.clinicaltrials.gov/large-docs/74/NCT02908074/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/74/NCT02908074/SAP_001.pdf